CLINICAL TRIAL: NCT00870025
Title: hCG Priming Prior to COH in Poor Responder IVF Patients
Brief Title: Human Chorionic Gonadotropin (hCG) Priming Prior to Controlled Ovarian Hyperstimulation (COH) in Poor Responder In Vitro Fertilization (IVF) Patients
Acronym: APPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVIMAD-LO-09-2008-01
Record Dates: First submitted 2008-10-25; First posted 2009-03-26 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Ovarian Response
Keywords: androgens; hCG; low response; IVF; Ovarian response in women with previous low response
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- hCG (Active Comparator): 200 IU rec hCG s.c./5 days, 4 doses prior to onset of COH
  Interventions: Biological: human chorionic gonadotropin; Biological: placebo
- placebo (Placebo Comparator): similar injection at same time points with similar diluent but no hCG
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: human chorionic gonadotropin — 200 IU, sc, every 5 days, 4 doses
  Arms: hCG
Biological: placebo — diluent, every 5 days, s.c., 4 doses

SUMMARY:
There is a decline in androgen concentration with ovarian aging. Also, ovarian response to COH in IVF cycles diminishes with ovarian aging. Recent evidence suggest that testosterone or DHEA may improve ovarian response in poor prognosis patients by increasing intraovarian androgen concentration. A physiological way to induce androgen synthesis within the ovary is to stimulate theca cells androgen production by hCG stimulation. By doing this in the previous cycle we might expect a better response to COH.

ELIGIBILITY:
Inclusion Criteria:

* previous IVF cycle with 5 or less mature follicles or 5 or less oocyte retrieved

Exclusion Criteria:

* 42 years or older
* BMI <18 or >30

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 2 weeks after intervention

SECONDARY OUTCOMES:
number of oocytes retrieved | 2 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Garcia-Velasco, MD, PhD, Principal Investigator — IVI Madrid
Locations (1):
- IVI-Madrid, Madrid, Spain

REFERENCES:
- [Background] Balasch J, Fabregues F, Penarrubia J, Carmona F, Casamitjana R, Creus M, Manau D, Casals G, Vanrell JA. Pretreatment with transdermal testosterone may improve ovarian response to gonadotrophins in poor-responder IVF patients with normal basal concentrations of FSH. Hum Reprod. 2006 Jul;21(7):1884-93. doi: 10.1093/humrep/del052. Epub 2006 Mar 3. PMID 16517559
- [Background] Massin N, Cedrin-Durnerin I, Coussieu C, Galey-Fontaine J, Wolf JP, Hugues JN. Effects of transdermal testosterone application on the ovarian response to FSH in poor responders undergoing assisted reproduction technique--a prospective, randomized, double-blind study. Hum Reprod. 2006 May;21(5):1204-11. doi: 10.1093/humrep/dei481. Epub 2006 Feb 13. PMID 16476678